CLINICAL TRIAL: NCT04792216
Title: Salmon Intake and Gut Health in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 20-1033
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Gut Microbiome; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wild Salmon (Experimental): Wild salmon fillets in a raw form
  Interventions: Other: Wild Salmon
- Farmed Salmon (Experimental): Farmed salmon fillets in a raw form
  Interventions: Other: Farmed Salmon

INTERVENTIONS:
Other: Wild Salmon — Wild salmon fillets
  Arms: Wild Salmon
Other: Farmed Salmon — Farm salmon fillets
  Arms: Farmed Salmon

SUMMARY:
The overall objective of this project is to determine the interplay of salmon as a whole food and its bioactive compound astaxanthin on gut microbiome, fecal metabolome, and inflammation in obese prediabetic individuals. Our central hypothesis is that dietary bioactive astaxanthin in the form of whole food salmon will effectively reduce inflammation in obese prediabetic individuals, and favorably change the gut microbiota composition and diversity. The investigators anticipate that these changes will result in improved metabolic outcomes in obesity and type 2 diabetes.

The two primary aims include:

Aim 1: Assess the anti-inflammatory effect of the salmon dietary intervention and the underlying mechanisms on the change in plasma levels of inflammatory cytokines important for the host immune response.

Aim 2: Identify whether the relationship between salmon consumption and decreased inflammation is mediated by the gut microbiome.

DETAILED DESCRIPTION:
The goal of this project is to determine whether increased intake of salmon as a whole food and its bioactive compound astaxanthin has a causal impact on preventing inflammation by promoting human gut microbiome homeostasis. Findings from this study will provide new insights into maintenance of gut microbiome and will inform effective dietary recommendations and interventions, thereby reducing inflammation-associated diseases in humans.

Aim: Evaluate the anti-inflammatory properties of astaxanthin-enriched salmon via re-balancing of human gut microbiome in obese prediabetic human subjects.

The investigators will use a randomized, double-blind, crossover feeding study with 15 obese prediabetic males and 15 obese prediabetic females (n=30) . Participants will consume two servings (3 oz per serving) of wild salmon (intervention 1) and farmed salmon (intervention 2) daily in random orders. Each intervention is 4 weeks long and the washout duration between the two interventions is 5 weeks. Primary outcomes will be determined by measuring the inflammatory response and gut microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant, non-lactating pre-menopausal females
* BMI 30-40 kg/m2
* Fasting blood glucose (without blood glucose-lowering drug) between 100-125 mg/dL
* Plasma total cholesterol ≤ 250 mg/dL, plasma triglyceride level ≤ 250 mg/Dl
* Age 30-50 years
* Weight stable over the last 3 months (< 2% body weight change)
* Sedentary and stable physical activity regimen 3 months prior (≤3 h/wk of moderate or high intensity exercise, resistance or aerobic training)
* Medication use stable for 6 months prior, and not include anti-inflammatory drugs (e.g. ibuprofen, aspirin)
* Not taking a carotenoid-containing or metabolism-altering supplement for the last 1 month, or have autoimmune diseases, and other malabsorptive disorders (including Crohn's, ileus or ulcerative colitis), liver or kidney insufficiency, allergies to tomatoes
* No current special diets or nutrient supplements, pre- or probiotics (~3 months)
* No tobacco smoking
* Limited consumption of alcoholic beverages ≤ 1/d
* No frequent habitual consumption of salmon or other astaxanthin-rich foods.

Exclusion Criteria:

* Pregnant, lactating, or menopausal females
* BMI < 30 or >40 kg/m2
* Fasting blood glucose <100 or >125 mg/dL; or taking blood glucose lowering medication
* Plasma total cholesterol >250 mg/dL, plasma triglyceride level >250 mg/Dl
* Age <30 or >50 years
* 2% body weight change over the last 3 months
* >3 h/wk of moderate or high intensity exercise, resistance or aerobic training for the 3 months prior
* Changing medications in the past 6 months
* Taking anti-inflammatory drugs (e.g. ibuprofen, aspirin), carotenoid-containing or metabolism-altering supplements (for the last 1 month), or have autoimmune diseases, and other malabsorptive disorders (including Crohn's, ileus or ulcerative colitis), liver or kidney insufficiency, or allergies to tomatoes
* Currently on a special diet or taking nutrient supplements, pre- or probiotics (~3 months)
* Tobacco smoking
* >1/d consumption of alcoholic beverages
* Frequent habitual consumption of salmon or other astaxanthin-rich foods.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Blood biomarkers/inflammatory cytokines | Over 32 weeks
  Blood from patients will be processed via centrifugation to archive plasma. A panel of 48 factors from Bio-Rad (Bio-Plex Pro™ Human Cytokine Screening Panel, 48-Plex #12007283) will be measured in plasma by Bio-Rad Bio-Plex analyzer. Five primary biomarkers (IL-1β, IL-6, IL-10, TNF-α, and MCP-1) will be confirmed by traditional ELISA
Gut Microbiome | Over 32 weeks
  Gut microbiota structure by 16S sequencing
Fecal metabolomics | Over 32 weeks
  Small molecules will be extracted using MTBE-based liquid:liquid extraction which results in lipid and aqueous fractions. Compounds will be "extracted" using commercial software (Mass Hunter, Agilent), quantitated using peak volumes and processed using Mass Profiler Professional (MPP, Agilent) to determine normalized compound intensities

SECONDARY OUTCOMES:
Urine Analysis | Over 32 weeks
  Urine samples will be collected for future metabolomics analysis. This analysis will generate a metabolomics profile in biospecimens, which will help us identify potential signatures related to salmon intake

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No